CLINICAL TRIAL: NCT01134133
Title: Can Hospital Acquired Pneumonia be Prevented in Patients Who Gurgle?
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow recruitment (preemptive treatment of gurglers, after association was published)
Sponsor: Bridgeport Hospital (Other)
Responsible Party: Constantine A. Manthous, MD, Bridgeport Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Gurgle
Record Dates: First submitted 2010-05-25; First posted 2010-05-31 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2010-02

CONDITIONS: Hospital Acquired Pneumonia in Gurgling Patients

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Anti-gurgling intervention — 1. head of bed 30 degrees or higher, 2. swallowing evaluation-based feeding, 3. sedatives titrated to minimal effective dose.

SUMMARY:
Hospital inpatients who have gurgling sounds heard during speech or breathing have been observed to have a higher risk of hospital acquired pneumonia. Patients who gurgle and who consent to participation will be randomized to receive routine clinical management or management to include measures employed to reduce risks of aspiration, namely, 1. head of bed up (30 degrees or higher), 2. swallowing evaluation by speech therapist (and feeding predicated on formal evaluation), 3. prompting managing physicians to reduce sedating medications to minimal effective dose.

ELIGIBILITY:
Inclusion Criteria:

* Gurglers who consent to participate

Exclusion Criteria:

* Non-gurglers
* Patients presenting with pneumonia prior to identification with gurgling
* Patients receiving comfort-care-only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Hospital acquired pneumonia | 14 days (average)